CLINICAL TRIAL: NCT02516930
Title: Crowdsourcing Versus Social Marketing Video Campaigns to Promote Condom Use: A Noninferiority Randomized Controlled Trial to Evaluate Promoting Condom Use Among MSM and Transgender Individuals in China
Brief Title: A Non-inferiority Randomized Controlled Trial to Evaluate Promoting Condom Use Among MSM and Transgender Individuals in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); SESH Global (Unknown); Guangdong Provincial Center for Dermatology and STD Control (Unknown); Shandong University (Other); Shandong Province Centers for Disease Control and Prevention (Other); University of California, San Francisco (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Joseph Tucker, MD, PhD, MA, Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 15-1522; 1R01AI114310-01 (NIH)
Record Dates: First submitted 2015-07-25; First posted 2015-08-06 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Human Immunodeficiency Virus; Sexually Transmitted Diseases
Keywords: health promotion; crowdsourcing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crowdsourced video (Other): One-minute crowd-sourced video promoting condom use among men who have sex with men and transgender individuals.
  Interventions: Behavioral: crowdsourced video
- Social marketing video (Other): One-minute social marketing video promoting condom use among men who have sex with men and transgender individuals
  Interventions: Behavioral: social marketing video

INTERVENTIONS:
Behavioral: crowdsourced video — video promoting condom use
  Arms: Crowdsourced video
Behavioral: social marketing video
  Arms: Social marketing video

SUMMARY:
This is a pragmatic, non-inferiority, randomized controlled trial comparing the effectiveness of two methods (crowdsourcing versus social marketing) for creating one-minute videos promoting condom use among MSM and TG in China. Crowdsourcing is the process of shifting individual tasks to a large group, often involving open contests and enabled through multisectoral partnerships.

DETAILED DESCRIPTION:
Crowdsourcing may be a powerful tool to spur the development of innovative videos to promote condom use among key populations such as men who have sex with men (MSM) and transgender (TG) individuals. The purpose of this randomized controlled trial is to compare the effect of a crowdsourced video and a social marketing video on condom use among Chinese MSM and TG who report condomless anal sex during the past three months. The crowdsourced video was developed using an open contest, formal transparent judging, and several prizes. The hypothesis is that a crowdsourced video will not be inferior (within a margin of 10%) to a social marketing video in terms of condomless sex at three to four weeks (with an additional follow-up at three months) of watching the video.

ELIGIBILITY:
Inclusion Criteria:

* The target population for the condom use substudy is males, 16 years of age or older, who were born biologically male or are transgender, have had condomless sex in the past three months and are willing to provide their cell mobile number.

Exclusion Criteria:

* Females

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1173 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Frequency of condomless sex following the assigned video intervention (3 wk) | 3 weeks following the video
  Frequency of men, defined as those who report condomless sex over the 3 week period divided by the total number of men who watched the video
Frequency of condomless sex following the assigned video intervention (3 month) | 3 months following the video
  Frequency of men, defined as those who report condomless sex over the 3 month period divided by the total number of men who watched the video

SECONDARY OUTCOMES:
Incremental cost | 3 weeks after baseline
  Incremental cost, defined as the cost associated with respective video interventions per individual who reported no sex or sex with a condom during the follow-up period.
Female condomless sex | 3 weeks and 3 months after baseline
  Frequency of men, defined as number of men who reported condomless vaginal or anal sex with a woman divided by the total number of men who viewed the video in that arm.
Male condomless sex | 3 weeks and 3 months after baseline
  Frequency of men, defined as number of men who reported condomless anal sex with a man divided by the total number of men who viewed the video in that arm.
Post-video condomless sex | 3 weeks after baseline
  Frequency of men, defined as number of men who reported condomless vaginal or anal sex with any partner immediately following the video intervention divided by the total number of men who viewed the video in that arm
Frequency of sex acts | 3 weeks and 3 months after baseline
  Frequency of men, defined as the number of men who had decreased total number of sex acts in the three weeks following the intervention compared to the three weeks immediately preceding the intervention in that arm
Condom self-efficacy | 3 weeks and 3 months after baseline
  Frequency of men, defined as number of men who had an increase in self-efficacy when comparing self-efficacy during the three weeks before baseline and the three weeks after the baseline, will measure again at 3 months and then compare baseline and three month data
Condom use social norms | 3 weeks and 3 months after baseline
  Frequency of men, defined as number of men who report higher levels of social norms when comparing their pre-intervention and post-intervention condom use norms.
Condom use negotiation | 3 weeks and 3 months after baseline
  Frequency of men, defined as the number of men who attempted to convince an unwilling partner to use a condom immediately following the video intervention divided by the total number of men who viewed the video in that arm
HIV testing | 3 weeks and 3 months after baseline
  Frequency of men, defined as the number of men who reported being tested for HIV during the interval between watching the video and following up compared to the number of men who followed up
STI testing | 3 weeks and 3 months after baseline
  Frequency of men, defined as the number of men who reported being tested for STIs (excluding HIV) during the interval between watching the video and following up compared to the number of men who followed up

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tucker, MD, PhD, MA, Principal Investigator — University of North Carolina
Locations (1):
- UNC Project-China, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Muessig KE, Bien CH, Wei C, Lo EJ, Yang M, Tucker JD, Yang L, Meng G, Hightow-Weidman LB. A mixed-methods study on the acceptability of using eHealth for HIV prevention and sexual health care among men who have sex with men in China. J Med Internet Res. 2015 Apr 21;17(4):e100. doi: 10.2196/jmir.3370. PMID 25900881
- [Background] Best J, Tang W, Zhang Y, Han L, Liu F, Huang S, Yang B, Wei C, Tucker JD. Sexual behaviors and HIV/syphilis testing among transgender individuals in China: implications for expanding HIV testing services. Sex Transm Dis. 2015 May;42(5):281-5. doi: 10.1097/OLQ.0000000000000269. PMID 25868142
- [Background] Bien CH, Muessig KE, Lee R, Lo EJ, Yang LG, Yang B, Peeling RW, Tucker JD. HIV and syphilis testing preferences among men who have sex with men in South China: a qualitative analysis to inform sexual health services. PLoS One. 2015 Apr 13;10(4):e0124161. doi: 10.1371/journal.pone.0124161. eCollection 2015. PMID 25875336
- [Background] Wei C, Muessig KE, Bien C, Yang L, Meng R, Han L, Yang M, Tucker JD. Strategies for promoting HIV testing uptake: willingness to receive couple-based and collective HIV testing among a cross-sectional online sample of men who have sex with men in China. Sex Transm Infect. 2014 Sep;90(6):469-74. doi: 10.1136/sextrans-2013-051460. Epub 2014 Apr 23. PMID 24760266
- [Background] Bien CH, Best JM, Muessig KE, Wei C, Han L, Tucker JD. Gay Apps for Seeking Sex Partners in China: Implications for MSM Sexual Health. AIDS Behav. 2015 Jun;19(6):941-6. doi: 10.1007/s10461-014-0994-6. PMID 25572834
- [Background] Han L, Bien CH, Wei C, Muessig KE, Yang M, Liu F, Yang L, Meng G, Emch ME, Tucker JD. HIV self-testing among online MSM in China: implications for expanding HIV testing among key populations. J Acquir Immune Defic Syndr. 2014 Oct 1;67(2):216-21. doi: 10.1097/QAI.0000000000000278. PMID 24991972
- [Background] Tucker JD, Muessig KE, Cui R, Bien CH, Lo EJ, Lee R, Wang K, Han L, Liu FY, Yang LG, Yang B, Larson H, Peeling RW. Organizational characteristics of HIV/syphilis testing services for men who have sex with men in South China: a social entrepreneurship analysis and implications for creating sustainable service models. BMC Infect Dis. 2014 Nov 25;14:601. doi: 10.1186/s12879-014-0601-5. PMID 25422065
- [Background] Tucker JD, Wei C, Pendse R, Lo YR. HIV self-testing among key populations: an implementation science approach to evaluating self-testing. J Virus Erad. 2015 Jan;1(1):38-42. doi: 10.1016/S2055-6640(20)31145-6. PMID 26005717
- [Background] Davis A, Best J, Luo J, Van Der Pol B, Dodge B, Meyerson B, Aalsma M, Wei C, Tucker JD; Social Entrepreneurship for Sexual Health Research Group. Differences in risk behaviours, HIV/STI testing and HIV/STI prevalence between men who have sex with men and men who have sex with both men and women in China. Int J STD AIDS. 2016 Sep;27(10):840-9. doi: 10.1177/0956462415596302. Epub 2015 Jul 15. PMID 26185041
- [Derived] Wang C, Tucker JD, Liu C, Zheng H, Tang W, Ling L. Condom use social norms and self-efficacy with different kinds of male partners among Chinese men who have sex with men: results from an online survey. BMC Public Health. 2018 Oct 16;18(1):1175. doi: 10.1186/s12889-018-6090-5. PMID 30326880
- [Derived] Liu C, Mao J, Wong T, Tang W, Tso LS, Tang S, Zhang Y, Zhang W, Qin Y, Chen Z, Ma W, Kang D, Li H, Liao M, Mollan K, Hudgens M, Bayus B, Huang S, Yang B, Wei C, Tucker JD. Comparing the effectiveness of a crowdsourced video and a social marketing video in promoting condom use among Chinese men who have sex with men: a study protocol. BMJ Open. 2016 Oct 3;6(10):e010755. doi: 10.1136/bmjopen-2015-010755. PMID 27697868
- See also: Social Entrepreneurship for Sexual Health Global — http://www.seshglobal.org
- See also: University of North Carolina website — http://www.unc.edu